CLINICAL TRIAL: NCT05818865
Title: "Principle Test" for Isolation and Characterization of Cancer Cells (CTC)-CXCR4+ Circulating in Belotero Loaded With CXCL12 in Patients With Solid Neoplasms (Endometrium, Kidney, Glioblastoma, Colorectal, Ovary and Lung).
Brief Title: "Principle Test" for Isolation and Characterization of Circulating Cancer Cells (CTC)-CXCR4+.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRAP4MET; 50/20 (Other: IRCCS I.N.T. "G. Pascale")
Record Dates: First submitted 2023-03-22; First posted 2023-04-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The development of an innovative device (CLG) consisting of an aqueous gel based on hyaluronic acid and commercially available (Belotero) able to be loaded and to release chemokine CXCL12 recreating a kind of "fake niche" able to attract immune cells- and CTCs-CXCR4+. The added value is the ability to attract and trap cells capable of leaking out and potentially with a higher metastatic capacity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- device (CLG) (Other): The development of an innovative device (CLG) consisting of an aqueous gel based on hyaluronic acid and commercially available (Belotero) able to be loaded and to release chemokine CXCL12 recreating a kind of "fake niche" able to attract immune cells- and CTCs-CXCR4+. The added value is the ability to attract and trap cells capable of leaking out and potentially with a higher metastatic capacity.
  Interventions: Device: CLG

INTERVENTIONS:
Device: CLG — The development of an innovative device (CLG) consisting of an aqueous gel based on hyaluronic acid and commercially available (Belotero) able to be loaded and to release chemokine CXCL12 recreating a kind of "fake niche" able to attract immune cells- and CTCs-CXCR4+. The added value is the ability to attract and trap cells capable of leaking out and potentially with a higher metastatic capacity.

SUMMARY:
This is multicentric, interventional, non farmacological and prospective study.

DETAILED DESCRIPTION:
The new CLG platform, a prototype owned by IRCCS Pascale Institute, is able to reconstruct a PMN for the capture of CTCs able to extravasare and colonize tissues at distance, a fundamental requirement to begin the process of metastasis formation. The purpose of the study is to evaluate in vitro the effectiveness of CLG in the isolation, recovery and subsequent molecular characterization of CTCs from peripheral blood of patients suffering from solid neoplasms (endometrium, kidney, colorectal, glioblastoma and lung).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Signature of Informed Consent
* Advanced solid neoplasm with metastases

Exclusion Criteria:

* Age <18
* Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
In vitro isolation of CTCs. | 2 years
  In vitro isolation of CTCs with high metastatic capacity from peripheral blood through CLG.Gene expression analysis will be performed using 250ng RNA for nCounter FLEX Analysis System (NanoStringTechnologies). Panels analyzed include the PanCancer Pathways and the PanCancer Progression. The data will be analyzed using the nSolver analysis software version 3.0
Real-Time PCR to evaluate the expression of Epithelium-Mesenchymal Markers | 2 years
  Expression analysis of Epithelium-Mesenchymal Markers (EPCAM, SNAIL, VIMENTIN, N-CADERIN, E-CADERIN) will be performed using Real-Time PCR.

SECONDARY OUTCOMES:
The correlation of the number and of biological/molecular characteristics of CTCs with the clinical/pathological characteristics of the patients in analysis and their prognosis. | 2 years
  The correlation of the number and of biological/molecular characteristics of CTCs with the clinical/pathological characteristics of the patients in analysis and their prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Portella, Principal Investigator — IRCCS I.N.T. "G. Pascale"
Locations (2):
- Italy (2):
  - Istitute Nazionale Tumori - Fondazione G. Pascale, Napoli
  - Istituto Nazionale Tumori - Fondazione "G.Pascale", IRCCS, Napoli